CLINICAL TRIAL: NCT03618706
Title: A Phase II Trial of Standard of Care Therapy With Involved Field Radiation Therapy for Selective Recurrent Ovarian Cancer
Brief Title: Standard of Care Therapy With Involved Field Radiation Therapy for Selective Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0299
Record Dates: First submitted 2018-07-09; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- involved-field RT + standard salvage treatment (Experimental): Patients receiving involved-field RT on recurred lesions + standard salvage treatment for recurrent ovarian cancer
  Interventions: Radiation: Involved-field radiotherapy

INTERVENTIONS:
Radiation: Involved-field radiotherapy — After the diagnosis of recurrences, patients will receive involved-field radiotherapy (gross tumor volume + margin) with any radiation dose scheme (≥45 Gy Biological Equivalent dose) as physician's discretion.

SUMMARY:
This study aims to investigate the effect of involved-field radiotherapy for recurrent ovarian cancer after primary standard treatment. We will investigate whether the addition of involved-field RT improves 2-year PFS in those patients than that of historical data (only with other standard salvage treatments as systemic chemotherapy ± maximum tumor resection).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed ovarian carcinoma
* Patients who received "standard treatment" for each stage as a primary treatment
* No. of recurrent lesions:

If, all in lung, or intra-abdominal or pelvis organs - ≤ 5 If, any in liver, bone, or spinal cord - ≤ 2

* Size of recurrent lesions ≤5 cm
* All recurrent lesions are available for involved-field radiotherapy
* Within 60 days before enrollment:
* Absolute neutrophil count ANC ≥ 500 / mm3
* Platelet ≥ 50,000 / mm3
* Hb ≥ 8.0 g / dl
* Good performance status (ECOG 0-1)

Exclusion Criteria:

* Brain metastasis
* Diffuse peritoneal carcinomatosis
* Malignant pleural effusion
* History of previous salvage radiotherapy for recurrent lesions
* History of other malignancy or severe/unstable medical condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2023-05-09 (Estimated); Study Completion 2023-05-09 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | 2 years after radiotherapy

SECONDARY OUTCOMES:
Local control of recurred lesions | 2 years after radiotherapy
Any other new recurrence events | 2 years after radiotherapy
Radiotherapy-related complications | 2 years after radiotherapy
Chemotherapy-free interval (The interval to delay the need for a new chemotherapy regimen for disease progression) | 2 years after radiotherapy
  It means the interval between the last date performing the previous chemotherapy (before the start of involved-field radiotherapy) and the first date performing the new regimen of chemotherapy (for the disease failures after the involve-field radiotherapy). We want to measure this interval because we want to check the capability of involved-field radiotherapy to delay the need for the new regimen of chemotherapy for the progressive diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No